CLINICAL TRIAL: NCT05472025
Title: Clinical Study of Combined Carotid Artery With Inferior Vena Cava Ultrasonography to Predict Hypotension After Induction of General Anesthesia: a Prospective Study
Brief Title: Clinical Study of Combined Carotid Artery With Inferior Vena Cava Ultrasonography to Predict Hypotension After Induction of General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Director, Tongji Hospital
Other Study IDs: TJ2022S073
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Ultrasound Guidance
Keywords: ultrasound; carotid artery; inferior vena cava; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Changes in blood pressure: Blood pressure assessment：The blood pressure and heart rate before induction and the blood pressure and heart rate per minute within 10 minutes after induction intubation were recorded. After induction of anesthesia, MAP < 60 mmHg, or the decrease rate exceeded 30% of the baseline value, was defined as the occurrence of hypotension

INTERVENTIONS:
Other:

SUMMARY:
Studies have shown that the clinical application of ultrasound to measure large blood vessels related parameters has been widely used to assess the blood volume status of patients, with the advantages of simple, non-invasive and non-radioactive, etc. However, these current methods using by ultrasound technology such as diameter and collapsibility index of the inferior vena cava parameters cannot fully reflect the blood volume, the sensitivity and specificity of predicting hypotension after induction are not very satisfied. Recent reports have demonstrated that respirophasic variation in carotid artery blood flow peak velocity (ΔVpeak) and carotid corrected flow time (FTc) can noninvasively assess patient responsiveness to fluids. Thus, we speculate that the combined measurement of the parameters of the carotid artery and the inferior vena cava may more comprehensively and accurately assess the patient's blood volume status, thereby accurately predicting the occurrence of hypotension after induction of anesthesia.

DETAILED DESCRIPTION:
Hypotension is common after induction of general anesthesia, with an incidence of 9% to 90%. Hypotension after induction of anesthesia may increase the risk of cardiovascular and cerebrovascular accidents, postoperative cognitive dysfunction, as well as increase the risk of postoperative acute myocardial injury and increase the mortality rate during hospitalization. The aim of this study is to establish an assessment method that can effectively predict hypotension after induction of anesthesia, so as to prevent possible harm to patients from perioperative hypotension. The study is planned to measure the peak flow velocity variation and corrected blood flow time of the carotid artery, the diameter and cross-sectional area of the inferior vena cava by applying ultrasound before anesthesia, and record the blood pressure and heart rate before induction of anesthesia, and the blood pressure and heart rate per minute within 10 minutes after induction of tracheal intubation. The mean arterial pressure (MAP) was recorded as the basal value before induction of anesthesia. After induction of anesthesia, MAP < 60 mmHg, or a decrease of more than 30% of the basal value, was defined as the occurrence of hypotension.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled to undergo surgery under general anesthesia
2. Age ≥ 18 years old
3. ASA I or II
4. The patient is clearly conscious and has the ability to cooperate with the ultrasound measurement
5. The patient signed the informed consent

Exclusion Criteria:

1. Emergency surgery
2. Consciousness disorder or mental disorder before surgery
3. Sudden emergency vital sign changes before surgery, life-threatening patients
4. Patients with preoperative respiratory distress, elevated intra-abdominal pressure, and expected difficult airway
5. Patients with preoperative autonomic nervous system disease
6. Patients with implantable pacemaker or cardioverter
7. Patients with preoperative peripheral vascular disease, severe cardiovascular disease, unstable angina or cardiac ejection fraction less than 40%
8. Pregnant women
9. Carotid artery stenosis
10. Severe carotid plaque

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Conscious adult patients with normal intra-abdominal pressure; no patients with severe diabetes, no severe carotid stenosis and plaque
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2022-10-26 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | Before induction of anesthesia
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | After induction of anesthesia to before tracheal intubation
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 1 minute
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 2 minute
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 3 minute
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 4 minute
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 5 minutes
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 6 minute
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 7 minutes
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 8 minutes
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 9 minutes
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography
Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography | after induction of anesthesia tracheal intubation 10 minutes
  Predictive power of the post-induced hypotension of combined carotid artery sonography with inferior vena cava sonography

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China